CLINICAL TRIAL: NCT00441207
Title: A Phase I Study of High-Dose IV Vitamin C Treatment in Patients With Solid Tumors
Brief Title: Study of High-Dose Intravenous (IV) Vitamin C Treatment in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Midwestern Regional Medical Center (Other)
Responsible Party: Principal Investigator, Chris Stephenson, DO, Midwestern Regional Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTCA 06-04; Ascorbic Acid Injection
Record Dates: First submitted 2007-02-26; First posted 2007-02-28 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Cancer
Keywords: IV Ascorbic Acid; IV Vitamin C; Cancer; Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Ascorbic Acid — Delivered via IV Infusion.

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of vitamin C (ascorbic acid) given by injection into the vein.

The second and third purpose of conducting this study is to observe any evidence of tumor response to the vitamin C and compare the level of fatigue (weakness), pain control, ability to do things, and quality of life, before and after vitamin C is given.

DETAILED DESCRIPTION:
Preclinical studies of pharmacologic doses of vitamin C (ascorbic acid, ascorbate) have shown significant anticancer effects in animal models and tissue culture investigations including cytotoxic effects in certain cancer cell lines at micromolar to millimolar concentrations.

Early clinical studies have shown that intravenous and oral doses of vitamin C may improve symptoms and prolong survival in terminal cancer patients. More recent double-blind placebo-controlled studies have shown that oral adminstration of vitamin C provides no benefit to cancer patients. Conversely, intravenous vitamin C administration raises plasma concentrations as high as 14 mM/L, and concentrations of 1-5 mM/L have been found to be selectively cytoxic to tumor cells in vitro.

The proposed Phase I trial with vitamin C should achieve millimolar concentrations of vitamin C that have been shown to kill tumor cells in vitro. The maximum tolerated dose (MTD), PK, possible drug accumulation with repeated dosing, quality of life, pain response, fatigue status, and hints of efficacy in patients with advanced cancer will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Primary histological diagnosis of advanced solid tumors (stage 3 and 4) and measurable disease.
* Disease must have progressed for which no available treatment provides clinical benefit.
* 18 years of age or older.
* No scheduled cancer therapy (chemotherapy, hormonal therapy, immune therapy, or radiation therapy) for three months after study entry, and the subject must have had their last therapy at least four (4) weeks prior to entry to this study.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Informed Consent - The patient must be willing and able to sign the informed consent prior to the start of the trial.
* Willingness to comply with the weekly phone calls between office visits.
* Willingness to undergo central line placement (e.g., port-a-catheter, central venous catheter, percutaneously inserted central catheter [PICC] line placement) and able to manage care of the entry site safely.
* Patients must be able to take food orally or have peg tube for feeding.
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Glucose-6-phosphate dehydrogenase deficiency (G6PD) (a relative contraindication)
* Renal insufficiency as evidenced by serum creatinine of ≥ 1.3 mg/dl or evidence of oxalosis by urinalysis.
* Chronic hemodialysis.
* Iron overload (a ferritin > 500 ng/ml).
* Wilson's disease.
* Compromised liver function with evidence of complete biliary obstruction or have a serum bilirubin of 2.0 or liver function tests (AST > 63, ALT > 95) exceeding 1.5 x the upper limit of normal.
* Pregnant or lactating female.
* Current tobacco use.
* Evidence of significant psychiatric disorder by history or examination that would prevent completion of the study or preclude informed consent.
* Aspirin use exceeding 325 mg per day.
* Acetaminophen use exceeding 2 g per day.
* Brain metastases that have not responded to therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of high dose IV vitamin C as a monotherapy | 1-1/2 years
Evaluate the pharmacokinetic profile of IV vitamin C at varying doses | 1-1/2 years

SECONDARY OUTCOMES:
Determine if vitamin C accumulates with repeated daily therapy by measuring peak and nadir levels | 1 year
Evaluate patient quality of life | Duration of Study
Observe patients for clinical and radiological evidence of anti-tumor activity at the end of treatment | Duration of Study

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Lis, Principal Investigator — Midwestern Regional Medical Center
Locations (1):
- CTCA @ Midwestern Regional Medical Center, Zion, Illinois, United States